CLINICAL TRIAL: NCT04386252
Title: Adaptive Phase I-II Clinical Trial of Preventive Vaccine Consisting of Autologous Dendritic Cells Previously Incubated With S-protein From Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2), in Subjects Negative for COVID-19 Infection and Anti-SARS-CoV-2 Antibodies
Brief Title: Phase I-II Trial of Dendritic Cell Vaccine to Prevent COVID-19 in Adults
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The FDA put our protocol on clinical hold and never gave an okay to start, so we decided not to proceed
Sponsor: Aivita Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CL-COV-P01-US
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — AV-COVID-19 vaccine; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Antigen Dose Exploration (Experimental): AV-COVID-19 consisting of autologous DC loaded with 0.1 mcg, 0.33 mcg or 1.0 mcg SARS-CoV-2 spike protein, with or without GM-CSF
  Interventions: Biological: AV-COVID-19
- Phase 2 (Experimental): Separate cohorts of patients who have 0 or >1 risk factor related to poor outcome for COVID-19 infection will receive AV-COVID-19 consisting of optimal antigen and GM-CSF formulation.
  Interventions: Biological: AV-COVID-19

INTERVENTIONS:
Biological: AV-COVID-19 — Autologous dendritic cells previously loaded ex vivo with SARS-CoV-2 spike protein
  Other Names: DC-ATA, DCV

SUMMARY:
This is an adaptive Phase I-II trial of a vaccine consisting of autologous dendritic cells previously loaded ex vivo with SARS-CoV-2 spike protein, with or without GM-CSF, to prevent COVID-19 in adults.

DETAILED DESCRIPTION:
Subjects eligible for treatment will be those who at baseline, are not actively infected with SARS-CoV-2, have no evidence of prior infection with SARS-CoV-2 based on serologic testing, and give informed consent for a vaccination with AV-COVID-19. The patient population will include the elderly and others at higher risk for poor outcomes after COVID-19 infection. For this reason, individuals will not be excluded solely on the basis of age, body mass index, history of hypertension, diabetes, cancer, or autoimmune disease.

After enrolling for screening, subjects will undergo a nasal swab test to exclude active COVID-19 infection and a rapid test for anti-coronavirus antibodies to exclude pre-existing anti-SARS-CoV-2 antibodies. 50 mL of blood will be collected, from which peripheral blood monocytes will be isolated and differentiated into DC before incubation with SARS-CoV-2 S-protein, during which time the protein is digested into 9 to 25 amino acid peptide sequences presented on the dendrites of DC in conjunction with histocompatibility class I and class II molecules. Safety and quality testing will be performed on a small quantity of the batch, and the remaining AV-COVID-19 will be cryopreserved for shipping to the treatment site.

Once the Study Drug is ready, if eligible, the subject will be seen at Study Week-0 for treatment. Prior to injection of the Study Drug, a nasal swab test will be collected to confirm that they are still negative for COVID-19, and blood will be drawn to determine baseline levels of anti-SARS-CoV-2 antibodies. At the treatment site, the product will be thawed and admixed with saline or (saline with GM-CSF), and within 5 hours of thawing, will be injected SC via a 25-gauge needle

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, in relatively good health with adequate physical and mental function, including factors associated with in increased risk for medical complications associated with COVID-19 infection or increased risk for exposure to SARS-CoV-2

Exclusion Criteria:

* Active COVID-19 infection by PCR testing, Pre-existing IgG or IgM SARS-CoV-2 antibodies, Pregnant, Known hypersensitivity to GM-CSF, Known active immune deficiency disease or active HIV, HBV, HCV, On active treatment with corticosteroids or other immunosupressive agent, Participated in previous COVID-19 vaccine study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Confirm safety | 1 year
  Confirm safety of AV-COVID-19 by adverse event monitoring

SECONDARY OUTCOMES:
Suggestion of efficacy | 1 month
  Measurement of IgG in subject blood
Optimal dose of SARS-CoV-2 antigen and GM-CSF | 1 months
  Measurement of IgG in subject blood

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Study Chair — AIVITA Biomedical